CLINICAL TRIAL: NCT00080600
Title: Central Motor Physiology in Polio Survivors
Brief Title: Brain Physiology in Polio Survivors
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040156; 04-N-0156
Record Dates: First submitted 2004-04-07; First posted 2004-04-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Postpoliomyelitis
Keywords: Post Polio Syndrome; Magnetic Stimulation; Fatigue; Exercise; Weakness; Transcranial Magnetic Stimulation; Post-Exercise Fatigue; Motor Neuron Disease; Cortical Reorganization; Intracortical Facilitation; Polio; Healthy Volunteer; HV
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Fatigue; Motor Activity; Asthenia; Motor Neuron Disease; Poliomyelitis

SUMMARY:
OBJECTIVE: Many persons who survive poliomyelitis develop pain, weakness, and fatigue many decades later. It is not known why some persons develop this syndrome and others do not. One possibility is that polio caused subclinical damage to the motor cortex. Autopsies in some polio patients have found damage to the brainstem and motor cortex as well as to spinal motor neurons. Alternatively, polio may have spared the motor cortex, but the cortex reorganized in different ways to compensate for the loss of spinal motor neurons. This study will first assess the integrity of central motor pathways in polio survivors with and without postpolio syndrome. The second goal will be to investigate differences in the intracortical mechanisms for controlling muscles affected and unaffected by polio.

STUDY POPULATION: 60 patients who survived polio in childhood. Only patients with an unequivocal history of polio will be referred to this study. Half of the patients will have the post-polio syndrome. 30 normal volunteers, aged 21-75.

DESIGN: Patients will be screened at the collaborating institution, the Uniformed Services University of the Health Sciences, which will also perform sensory evoked potential testing and MRI. At NIH, motor evoked potentials will be elicited from all four limbs using transcranial magnetic stimulation to assess central motor conduction time and threshold. Intracortical facilitation will be used to assess using paired-pulse magnetic stimulation. Two muscles will be tested in each patient, one affected by polio and one unaffected by polio. In the affected muscle, intracortical facilitation will be assessed again after exercises it until it fatigues.

OUTCOME PARAMETERS: Cortical thresholds and central motor conduction times to all four limbs will be measured in patients and compared to normal subjects. The mean intracortical facilitation at rest will be compared in affected and unaffected muscles in polio patients with and without post-polio syndrome.

DETAILED DESCRIPTION:
OBJECTIVE: Many persons who survive poliomyelitis develop pain, weakness, and fatigue many decades later. It is not known why some persons develop this syndrome and others do not. One possibility is that polio caused subclinical damage to the motor cortex. Autopsies in some polio patients have found damage to the brainstem and motor cortex as well as to spinal motor neurons. Alternatively, polio may have spared the motor cortex, but the cortex reorganized in different ways to compensate for the loss of spinal motor neurons. This study will first assess the integrity of central motor pathways in polio survivors with and without postpolio syndrome. The second goal will be to investigate differences in the intracortical mechanisms for controlling muscles affected and unaffected by polio.

STUDY POPULATION: 60 patients who survived polio in childhood. Only patients with an unequivocal history of polio will be referred to this study. Half of the patients will have the post-polio syndrome. 30 normal volunteers, aged 21-80.

DESIGN: Patients will be screened at the collaborating institution, the Uniformed Services University of the Health Sciences, which will also perform sensory evoked potential testing. At NIH, motor evoked potentials will be elicited from all four limbs using transcranial magnetic stimulation to assess central motor conduction time and threshold. MRI scans of the brain or spine will be performed in patients with abnormal evoked potentials. Intracortical facilitation will be assessed using paired-pulse magnetic stimulation. Two muscles will be tested in each patient, one affected by polio and one unaffected by polio. In the affected muscle, intracortical facilitation will be assessed again after exercises it until it fatigues.

OUTCOME PARAMETERS: Cortical thresholds and central motor conduction times to all four limbs will be measured in patients and compared to normal subjects. The mean intracortical facilitation at rest will be compared in affected and unaffected muscles in polio patients with and without post-polio syndrome.

ELIGIBILITY:
* INCLUSION CRITERIA:

POLIO PATIENTS:

Complete screening evaluation.

Meet clinical criteria for diagnosis of past polio (see below).

Meet clinical criteria for the diagnosis of PPS (PPS group only) and have new muscle weakness.

Age 21 or older.

CLINICAL CRITERIA FOR PAST POLIO (CONFIRMED):

Clinically compatible signs and symptoms of paralytic poliomyelitis (acute flaccid paralysis of one or more limbs).

Decreased or absent tendon reflexes on the affected limbs.

No persistent sensory or cognitive loss.

No other apparent cause (including laboratory investigation to rule out other causes of similar syndrome).

Neurological deficit present 60 days after onset of initial symptoms.

Associated with isolation of either vaccine or wild poliovirus from a clinical specimen.

CLINICAL CRITERIA FOR POST-POLIO SYNDROME:

History of polio with partial or complete neurological and functional recovery.

Stable function greater than 15 years.

New onset of one or more of the following: fatigue, weakness, atrophy, muscle pain, functional loss.

Exclusion of other explanations for the symptomatology.

Neurological evaluation demonstrating: lower motor neuron dysfunction (confirmed by EMG, imaging studies or muscle biopsy), no sensory loss.

Must have new onset of muscle weakness in one or more limb muscles, as determined by history and clinical examination.

NORMAL VOLUNTEERS:

Healthy adult volunteers ages 21-80 who are willing to participate.

EXCLUSION CRITERIA:

Neurological diseases or conditions, other than polio, that in the judgment of the investigators may account for the symptoms or interfere with the experimental interventions.

Implanted devices, such as pumps, pacemakers, or metal fragments in the skull or eye.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-04-06; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Cashman NR, Maselli R, Wollmann RL, Roos R, Simon R, Antel JP. Post-poliomyelitis syndrome: evidence of ongoing denervation in symptomatic and asymptomatic patients. Birth Defects Orig Artic Ser. 1987;23(4):237-9. No abstract available. PMID 3620621
- [Derived] Prokhorenko OA, Vasconcelos OM, Lupu VD, Campbell WW, Jabbari B. Sensory physiology assessed by evoked potentials in survivors of poliomyelitis. Muscle Nerve. 2008 Oct;38(4):1266-71. doi: 10.1002/mus.21093. PMID 18816600
- [Derived] Lupu VD, Danielian L, Johnsen JA, Vasconcelos OM, Prokhorenko OA, Jabbari B, Campbell WW, Floeter MK. Physiology of the motor cortex in polio survivors. Muscle Nerve. 2008 Feb;37(2):177-82. doi: 10.1002/mus.20913. PMID 17990291